CLINICAL TRIAL: NCT05591274
Title: Modulating Intraoperative Vasectomy Pain Using the SmileyScope Virtual Reality Interface
Brief Title: Virtual Reality Technology for Vasectomy Pain Modulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20220880
Record Dates: First submitted 2022-10-17; First posted 2022-10-24 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Vasectomy; Pain, Postoperative; Anxiety Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into one of three groups (interactive virtual reality, static virtual reality, and no virtual reality).
Masking Description: Patients will be randomized into one of three groups (interactive virtual reality, static virtual reality, and no virtual reality). Randomization sequence will be generated using a validated random number generator, and allocation concealment will be achieved via opaque envelope. Treatment (vasectomy with interactive VR, vasectomy with static VR, or vasectomy with no VR) will be known to patient and care provider only once the vasectomy procedure begins.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Interactive VR (Experimental): Patients will be wearing a virtual reality headset preloaded with an interactive VR scenario.
  Interventions: Device: SmileyScope Virtual Reality Headset
- Static VR (Experimental): Patients will be wearing a virtual reality headset preloaded with a static, non-interactive VR scenario.
  Interventions: Device: SmileyScope Virtual Reality Headset
- Control (No Intervention): Patients will not be wearing any virtual reality headset.

INTERVENTIONS:
Device: SmileyScope Virtual Reality Headset — The SmileyScope Virtual Reality Headset is a VR headset undergoing study for approval by the U.S. Food and Drug Administration (FDA) to reduce pain and anxiety in patients aged 4 years and older undergoing needle blood draw or injection procedures. Currently, this device has been granted entrance to the FDA Safer Technologies Program. The device comes pre-loaded with either an interactive or static virtual reality scenario.
  Arms: Interactive VR; Static VR

SUMMARY:
This study will evaluate whether or not wearing a virtual reality (VR) headset reduces pain and anxiety in patients undergoing vasectomy. The headset being used is the SmileyScope virtual reality interface, a device already undergoing study for approval by the U.S. Food and Drug Administration (FDA) to reduce pain and anxiety in patients aged 4 years and older undergoing needle blood draw or injection procedures. In this study, the SmileyScope virtual reality interface is considered an investigational device because it is not yet approved for use in adult males undergoing vasectomy.

DETAILED DESCRIPTION:
Vasectomy is a safe and effective procedure for permanent sterilization in males. More than 500,000 vasectomies are performed annually in the United States, and that number is expected to grow rapidly in the coming years. The procedure is safe and can be quickly performed in an outpatient setting. Complications of vasectomy are rare, and can include hematoma and infection, spermatic granulomas, and post-vasectomy pain syndrome in rare cases. Like all outpatient surgical procedures where the patient is not under general anesthesia, vasectomies involve intraoperative and immediate post-operative pain. While use of the no-scalpel technique and local anesthetic reduces intraoperative pain, expected operative pain is still one of the main reasons patients cite for not undergoing the procedure.

In our current study, the investigators aim to further modulate intraoperative pain using virtual reality goggles. In clinical trials, the SmileyScope device has been shown to reduce procedural pain in the pediatric population during venipuncture or intravenous cannulation. Results from those studies showed a statistically significant reduction in pain during intravenous procedures in the emergency department. This VR headset is undergoing study for approval by the U.S. Food and Drug Administration (FDA) to reduce pain and anxiety in patients aged 4 years and older undergoing needle blood draw or injection procedures. Currently, this device has been granted entrance to the FDA Safer Technologies Program. In this study, the SmileyScope virtual reality interface is considered an investigational device because it is not yet approved for use in adult males undergoing vasectomy. The aim of this study is to investigate whether this same virtual reality modality can be utilized to reduce pain during vasectomies.

ELIGIBILITY:
Inclusion Criteria:

* Adult males 18 years or older who are undergoing elective vasectomy

Exclusion Criteria:

* Have a serious comorbid illness or condition that, in the opinion of the investigator, may compromise the safety or compliance of the subject or preclude successful completion of the study
* History of chronic pain disorder or chronic narcotic use
* Significant refractive error, unilateral blindness, epilepsy, or other conditions such as skin infections, cancer, etc. which could compromise the physical function of the headset.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhan Qureshi, PhD, Principal Investigator — University of Miami
Locations (1):
- Desai Sethi Urology Institute, University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Interactive Virtual Reality (VR): Patients will be wearing a virtual reality (VR) headset preloaded with an interactive VR scenario.
  SmileyScope Virtual Reality Headset: The SmileyScope Virtual Reality Headset is a VR headset undergoing study for approval by the U.S. Food and Drug Administration (FDA) to reduce pain and anxiety in patients aged 4 years and older undergoing needle blood draw or injection procedures. Currently, this device has been granted entrance to the FDA Safer Technologies Program. The device comes pre-loaded with either an interactive or static virtual reality scenario.
- Static Virtual Reality (VR): Patients will be wearing a virtual reality headset preloaded with a static, non-interactive VR scenario.
  SmileyScope Virtual Reality Headset: The SmileyScope Virtual Reality Headset is a VR headset undergoing study for approval by the U.S. Food and Drug Administration (FDA) to reduce pain and anxiety in patients aged 4 years and older undergoing needle blood draw or injection procedures. Currently, this device has been granted entrance to the FDA Safer Technologies Program. The device comes pre-loaded with either an interactive or static virtual reality scenario.
Period: Overall Study
Arm/Group | Interactive Virtual Reality (VR) | Static Virtual Reality (VR) | Control
Started | 40 | 40 | 40
Completed | 40 | 40 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interactive VR | Static VR | Control | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.33 (7.32) | 40.58 (4.92) | 40.13 (4.72) | 40.01 (5.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 40 | 40 | 40 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 25 | 23 | 76
  Not Hispanic or Latino | 10 | 15 | 16 | 41
  Unknown or Not Reported | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 5 | 11
  White | 36 | 32 | 31 | 99
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pre-operative Anxiety
Description: Anxiety will be measured via the State-Trait Anxiety Inventory (STAI) anxiety score [Range 20-80; 20 = low anxiety, 80 = high anxiety]
Time Frame: up to 1 day
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Interactive VR | Static VR | Control
Number analyzed (Participants) | 40 | 40 | 40
score on a scale | 14 [12 to 15] | 13.5 [13 to 15] | 14 [12 to 15]

2. Primary Outcome: Post-operative Anxiety
Description: as for outcome 1
Time Frame: up to 1 day
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Interactive VR | Static VR | Control
Number analyzed (Participants) | 40 | 40 | 40
score on a scale | 14.5 [13 to 15] | 14 [13 to 15] | 15 [13 to 15]

3. Primary Outcome: Subjective Pre-operative Pain
Description: Pain will be measured via numeric Likert pain scale [0-10; 0 = no pain, 10 = highest pain]
Time Frame: up to 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interactive VR | Static VR | Control
Number analyzed (Participants) | 40 | 40 | 40
score on a scale | 0.05 (0.32) | 0 (0) | 0.05 (0.316)

4. Primary Outcome: Subjective Post-operative Pain
Description: Pain will be measured via numeric Likert pain scale; compared to baseline pain scale in pre-operative period [0-10; 0 = no pain, 10 = highest pain]
Time Frame: up to 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interactive VR | Static VR | Control
Number analyzed (Participants) | 40 | 40 | 40
score on a scale | 2.875 (1.571) | 2.447 (1.554) | 2.325 (1.623)

5. Primary Outcome: Post-procedure Satisfaction
Description: Satisfaction will be measured via a questionnaire scored by Likert scale. Questionnaire will ask:
  "How satisfied were you with today's procedure, with 0 being not satisfied at all, and 10 being the most satisfied?" "How helpful was VR in managing your vasectomy today" (0 is least helpful, 10 is most helpful)"
Time Frame: up to 1 day
Population: Only Participants randomized to one of the two VR arms were asked to complete the post procedure satisfaction survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interactive VR | Static VR | Control
Number analyzed (Participants) | 40 | 40 | 40
score on a scale
  How satisfied were you with today's procedure? (0 not satisfied at all; 10 most satisfied) | 4.86 (0.42) | 4.92 (0.28) | 4.61 (1.02)
  How helpful was VR in managing your vasectomy today? (0 least helpful, 10 most helpful): number analyzed (Participants) | 40 | 40 | 0
  How helpful was VR in managing your vasectomy today? (0 least helpful, 10 most helpful) | 3.92 (1.3) | 4.06 (1.04) |

6. Secondary Outcome: Physiological Intra-operative Heart Rate
Description: Heart rate will be measured intra-operatively using a FitBit Versa 3 device worn on the patient's wrist.
Time Frame: up to 1 day
Measure: Mean (Standard Deviation); unit: beats per minute (BPM)
Groups:
- Interactive Virtual Reality (VR): Patients will be wearing a virtual reality headset preloaded with an interactive VR scenario.
  SmileyScope Virtual Reality Headset: The SmileyScope Virtual Reality Headset is a VR headset undergoing study for approval by the U.S. Food and Drug Administration (FDA) to reduce pain and anxiety in patients aged 4 years and older undergoing needle blood draw or injection procedures. Currently, this device has been granted entrance to the FDA Safer Technologies Program. The device comes pre-loaded with either an interactive or static virtual reality scenario.
Arm/Group | Interactive Virtual Reality (VR) | Static Virtual Reality (VR) | Control
Number analyzed (Participants) | 40 | 40 | 40
beats per minute (BPM) | 77.8 (13.5) | 75.2 (10.9) | 77.2 (12.1)

7. Secondary Outcome: Physiological Intra-operative Oxygen Saturation
Description: Oxygen saturation will be measured intra-operatively using a FitBit Versa 3 device worn on the patient's wrist.
Time Frame: up to 1 day
Population: Data was not collected due to an oversight in the study design. All vital sign parameters were planned to be collected via FitBit Versa 8. However, once the research team realized it was not possible to capture oxygen saturation and temperature with this device, the protocol should have been amended. A Note-to-File was created to document this protocol deviation.
Arm/Group | Interactive VR | Static VR | Control
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Physiological Intra-operative Skin Temperature
Description: Skin temperature will be measured intra-operatively using a FitBit Versa 3 device worn on the patient's wrist.
Time Frame: up to 1 day
Population: as for outcome 7
Arm/Group | Interactive VR | Static VR | Control
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Physiological Post-operative Heart Rate
Description: Heart rate will be measured post-operatively using a FitBit Versa 3 device worn on the patient's wrist.
Time Frame: up to 1 day
Measure: Mean (Standard Deviation); unit: beats per minute (BPM)
Arm/Group | Interactive Virtual Reality (VR) | Static Virtual Reality (VR) | Control
Number analyzed (Participants) | 40 | 40 | 40
beats per minute (BPM) | 75.9 (12.2) | 75.9 (12.2) | 75.1 (13.9)

10. Secondary Outcome: Physiological Post-operative Oxygen Saturation
Description: Oxygen saturation will be measured post-operatively using a FitBit Versa 3 device worn on the patient's wrist.
Time Frame: up to 1 day
Population: as for outcome 7
Arm/Group | Interactive VR | Static VR | Control
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Physiological Post-operative Skin Temperature
Description: Skin temperature will be measured post-operatively using a FitBit Versa 3 device worn on the patient's wrist.
Time Frame: up to 1 day
Population: as for outcome 7
Arm/Group | Interactive VR | Static VR | Control
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 Day
Description: Adverse Events (AEs) were collected only on the day of procedure (day of vasectomy)
Arm/Group | Interactive VR | Static VR | Control
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 1/40 | 0/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interactive VR (N=40) | Static VR (N=40) | Control (N=40)
Vasovagal Reaction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT05591274/Prot_SAP_000.pdf